CLINICAL TRIAL: NCT02103959
Title: A Prospective, Comparative, Randomized, Multi-Center, Double-Blinded, Placebo-Controlled, Phase 2a Study of the Safety and Efficacy of CMX-2043 for Periprocedural Injury Protection in Subjects Undergoing Coronary Angiography at Risk of Radio-contrast Induced Nephropathy (CARIN)
Brief Title: Safety and Efficacy of CMX-2043 for Protection of the Heart and Kidneys in Subjects Undergoing Coronary Angiography
Acronym: CARIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ischemix, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMX-2043-2aK
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2014-06

CONDITIONS: Non STEMI; Unstable Angina
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable | interventions — alpha-N-(1,2-dithiolane-3-pentanoyl)glutamylalanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CMX-2043 2.4 mg/Kg (Experimental): Bolus injection of investigational product given prior to the cardiac catheterization and placebo given 24 hours after the first dose.
  Interventions: Drug: CMX-2043
- CMX-2043 3.6 mg/kg (Experimental): Bolus injection of investigational product given prior to the cardiac catheterization and placebo given 24 hours after the first dose.
  Interventions: Drug: CMX-2043
- CMX-2043 2.4 mg/kg given twice (Experimental): Bolus injection of investigational product given prior to the cardiac catheterization and again 24 hours after the first dose.
  Interventions: Drug: CMX-2043
- Placebo comparator (Placebo Comparator): Placebo comparator (PBS) given prior to cardiac catheterization and again 24 hours after the first dose.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: CMX-2043 — Slow bolus IV administration of CMX-2043
  Arms: CMX-2043 2.4 mg/Kg; CMX-2043 2.4 mg/kg given twice; CMX-2043 3.6 mg/kg
Drug: Placebo comparator — Slow bolus IV administration of PBS
  Arms: Placebo comparator

SUMMARY:
The objective of this study is to evaluate CMX-2043 for prevention of renal and cardiac injury associated with coronary angiography in patients with acute coronary syndrome (ACS), but excluding ST-elevation myocardial infarction (STEMI) patients. This study will specifically examine the ability of CMX-2043 to prevent acute renal injury following coronary angiography. The study will also examine the ability of CMX 2043 for prevention of periprocedural cardiac injury. Information will be obtained relating to the ability of CMX 2043 for prevention of major adverse cardiac and renal events following the procedure. Additional information will be obtained in this study to evaluate safety of the drug. Dose and regimen information will also be obtained for future clinical studies of CMX-2043.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age.
2. Subjects with acute coronary syndrome (excluding STEMI).
3. Subjects undergoing coronary angiography with the possibility of going on to PCI. However, if it is known that the patient is unlikely to undergo PCI, the patient should not be enrolled.
4. Subjects must meet either one of the following criteria:

   1. An eGFR < 45 mL/min as determined by the MDRD equation
   2. An eGFR < 60 mL/min as determined by the MDRD equation and at least one of the following:

   i. Over 75 years of age ii. Diabetes mellitus iii. Ejection fraction less than 40% iv. Hypotension v. Congestive heart failure (NYHA stage II or higher) vi. Anemia (hemoglobin below 10 g/dL at screening)
5. Female subjects must also meet any one of the following criteria:

   1. Surgically sterile with bilateral tubal ligation or hysterectomy
   2. Post-menopausal for at least one year
   3. If of child-bearing potential, practicing an acceptable method of birth control for the duration of the study as judged by the investigator, such as condoms, foams, jellies, diaphragm, intrauterine device or abstinence.
6. Subjects free of non-cardiac acute injuries or illnesses that, in the opinion of the investigator, could put the subject at risk or obscure the interpretation of results.
7. Subjects willing to undergo pre-and post-study blood and urine collection, physical exams and laboratory investigations.
8. Subjects willing to provide signed written informed consent form.

Exclusion Criteria:

1. Subjects undergoing elective coronary angiography (i.e., stable angina).
2. Subjects with end-stage renal disease (i.e., eGFR < 15).
3. Subjects with ST-elevation myocardial infarction (STEMI)
4. Subjects who experienced cardiac arrest associated with the current admission which required chest compressions or cardiopulmonary resuscitation.
5. Subjects who experienced a life threatening arrhythmia associated with the current admission such as ventricular fibrillation or ventricular tachycardia.
6. Subjects who weigh over 125 kg.
7. Subjects with an active history of psychiatric disorders likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements.
8. Subjects with a history of alcohol or drug abuse within one year of screening.
9. Subjects with uncorrected clinically significant abnormalities of clinical laboratory tests which in the investigators opinion will interfere with the study conduct.
10. Subjects with non-cardiac acute illness or injuries in which the investigator considers will increase the risk to the subject or to the study's success or which will obscure the interpretation of the results.
11. Subject with chronic diseases considered by the investigator unfit for the procedure or which will increase the risk to the subject or to the study's success or which will obscure the interpretation of results.
12. Subjects who are currently enrolled or who have participated in a clinical study within 30 days of screening or within 5 half-lives of another study drug, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prevention of acute kidney injury (AKI). | Three days
  Reduction in the incidence of AKI as determined by the KDIGO definition of AKI compared to placebo.

SECONDARY OUTCOMES:
Reduction in biomarkers of AKI | Three days
  Reduction in renal injury as determined by renal biomarkers in the treatment groups compared to placebo.
Trends in clinical outcomes | 90 days
  Incidence of major adverse cardiac events (MACE) or major adverse kidney events (MAKE) or other clinical complications in the treatment groups compared to placebo.
Prevention of cardiac injury in unstable angina (UA) subjects who go on to PCI. | Three days
  Reduction in cardiac injury as determined by cardiac biomarkers in the treatment groups compared to placebo
Safety monitoring | 90 days
  Assessments of treatment emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Lader, PhD, Study Director — Ischemix, LLC